CLINICAL TRIAL: NCT03065504
Title: Pilot Study on the Effects of Oral Turmeric and Turmeric-containing Tablets on Sebum Production
Brief Title: Turmeric and Turmeric-containing Tablets and Sebum Production
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 948358
Record Dates: First submitted 2016-11-01; First posted 2017-02-28 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Skin Inflammation
MeSH Terms: conditions — Dermatitis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Turmeric group (Active Comparator): 2,000 mg turmeric per day - supplied by Banyan® Botanicals )
  o Each tablet contains 500 mg of Turmeric (Curcuma longa). Subjects will take 2 tablets twice per day, with a total daily dose of 2,000 mg.
  Interventions: Dietary Supplement: Turmeric
- Turmeric-containing combination tablets (Active Comparator): • 2,000 mg Healthy Skin™ Tablets, contains:
  * Turmeric (Curcuma longa) - 50 mg/tablet
  * Hemidesmus Indicus root (Anantamul)
  * Indian Madder root
  * Neem leaf
  * Gotu Kola leaf
  * Indian TInospora stem
  * Amla fruit
  * Licorice root
  * Phyllanthus Amarus herb Each tablet contains 500mg total of the above herbs. There is 50 mg of Turmeric in each Healthy Skin ™ tablet. Subjects will take 2 tablets twice per day, which will be a total daily dose of 200 mg of Turmeric. This is comparable to the daily amount of Turmeric in many commercially-available Turmeric supplements; therefore, it is valuable to compare this formulation to the turmeric-only tablets.
  Interventions: Dietary Supplement: Turmeric-containing combination tablet
- Placebo tablets group (Placebo Comparator): * Supplement appearing similar to those in the turmeric and curcumin groups, supplied by Banyan® Botanicals
  * Ingredients (all organic): Placebo ingredients: Rice hulls concentrate, Maltodextrin, Micro Crystalline Cellulose, Beet Root Powder, Dutch coco powder
  * Dose: subjects in this group will take 2 tablets twice per day
  Interventions: Dietary Supplement: Placebo tablets

INTERVENTIONS:
Dietary Supplement: Turmeric
  Arms: Turmeric group
Dietary Supplement: Turmeric-containing combination tablet
  Arms: Turmeric-containing combination tablets
Dietary Supplement: Placebo tablets
  Arms: Placebo tablets group

SUMMARY:
A noticeably increasing number of patients are asking for naturally based extracts and ingredients as supplementary dermatologic remedies. Patients are seeking natural and cost-effective skin care alternatives in place of prescription medications and procedures. This study will isolate the effects of oral turmeric and assess a combination tablet that includes turmeric on sebum production in healthy subjects.

DETAILED DESCRIPTION:
Turmeric (Curcuma longa) is a spice that has been shown to exhibit anti-inflammatory, antimicrobial, antioxidant, anti-neoplastic properties, and even potential to improve mental illnesses. In western herbalism, Turmeric is primarily used as an anti-inflammatory agent. In India, turmeric is used in Ayurvedic medicine for the treatment of acne. It has been used both internally and externally.

Curcumin is a phytochemical derived from turmeric and believed to be one of the key active components of turmeric. Curcumin is reported to have activity as an antibacterial and anti-inflammatory agent and has been used as a paste for skin eruptions and infections. Previous basic science work by Dr. Raja Sivamani's lab has shown that both turmeric and curcumin inhibit lipid synthesis in human sebocytes, the cells responsible for the production of sebum

The goal of this study is to evaluate how ingestion of turmeric and tablets that have a combination of herbs including turmeric may modulate sebum production.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50 years of age, and
2. Subject must be able to read and comprehend study procedures and consent forms.

Exclusion Criteria:

1. Subject should be generally healthy and have no smoking history in the past one year, and must have no history of diabetes, metabolic syndrome, known cardiovascular disease, malignancy, kidney disease, or chronic steroid use.
2. Subjects who consume more than 6 servings of caffeine per day, such as coffee and energy drinks (example - Red Bull).
3. Subjects with known allergies to herbal ingredients.
4. Subjects with known EKG changes.
5. Those who used topical medications in the past two weeks or systemic antibiotics within one month of starting the study.
6. Subjects who are postmenopausal
7. Those who are pregnant or breastfeeding.
8. Those that are prisoners or cognitively impaired.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-11; Primary Completion 2017-08-28 (Actual); Study Completion 2017-08-28 (Actual)

PRIMARY OUTCOMES:
Change in facial Sebum production at 4 weeks | 4 weeks
  The investigators will use Sebutapes placed on the forehead to measure facial sebum production for 60 minutes at baseline and after 4 weeks. The tapes will collect the facial sebum produced during that time.

SECONDARY OUTCOMES:
Change from baseline in sebum profile, such as inflammatory markers, at 4 weeks | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, M.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Dermatology Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thangapazham RL, Sharma A, Maheshwari RK. Beneficial role of curcumin in skin diseases. Adv Exp Med Biol. 2007;595:343-57. doi: 10.1007/978-0-387-46401-5_15. PMID 17569219
- [Background] Chainani-Wu N. Safety and anti-inflammatory activity of curcumin: a component of tumeric (Curcuma longa). J Altern Complement Med. 2003 Feb;9(1):161-8. doi: 10.1089/107555303321223035. PMID 12676044
- [Derived] Vaughn AR, Pourang A, Clark AK, Burney W, Sivamani RK. Dietary supplementation with turmeric polyherbal formulation decreases facial redness: a randomized double-blind controlled pilot study. J Integr Med. 2019 Jan;17(1):20-23. doi: 10.1016/j.joim.2018.11.004. Epub 2018 Nov 22. PMID 30527287